CLINICAL TRIAL: NCT02529124
Title: An Investigation of the the Effect of Nutrient Support, or Nutrient Plus Physical Activity on Musculoskeletal Health and Function in Men and Women Aged 55 to 70 Years
Brief Title: Nutrient Support to Body Composition and Healthy Ageing
Acronym: BCHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phil Jakeman (Other)
Responsible Party: Sponsor-Investigator, Phil Jakeman, Phil Jakeman, University of Limerick
Organization: University of Limerick (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: EHSREC10_45
Record Dates: First submitted 2015-08-12; First posted 2015-08-19 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Sarcopenia; Osteopenia
Keywords: Ageing; Body Composition; Nutrition; Physical Activity
MeSH Terms: conditions — Sarcopenia; Bone Diseases, Metabolic; Motor Activity | interventions — maltodextrin; Proteins; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CONTROL (Placebo Comparator): a group of subjects receiving a placebo nutrient supplement (per kg of body mass: 0.25g maltodextrin; energy ~ 160 kcal per day) in two equal portions at the two low protein meals of the day, i.e. breakfast and lunch every day for a period of 24 weeks
  Interventions: Dietary Supplement: CONTROL
- PROTEIN (Active Comparator): a group of subjects receiving a nutrient supplement (per kg of body mass: 0.33g milk protein + 0.25ug vitamin D + 10mg calcium; energy ~ 160 kcal per day) in two equal portions at the two low protein meals of the day, i.e. breakfast and lunch every day for a period of 24 weeks
  Interventions: Dietary Supplement: PROTEIN
- PROTEIN+PHYSICAL ACTIVITY (Active Comparator): a group of subjects receiving a nutrient supplement (per kg of body mass: 0.33g milk protein + 0.25ug vitamin D + 10mg calcium; energy ~ 160 kcal per day) in two equal portions at the two low protein meals of the day, i.e. breakfast and lunch every day for a period of 24 weeks plus a prescribed regimen of physical activity
  Interventions: Dietary Supplement: PROTEIN; Behavioral: PHYSICAL ACTIVITY

INTERVENTIONS:
Dietary Supplement: CONTROL — Maltodextrin (generic) in powder form, flavoured and instantised to be dissolved in water.
  Other Names: MALTODEXTRIN
  Arms: CONTROL
Dietary Supplement: PROTEIN — The milk protein matrix (PROTEIN) comprised a 9:2:1 ratio of milk protein concentrate (MPC, 80% (w/w protein) Glanbia Nutritionals, Kilkenny, Ireland), whey protein concentrate hydrolysate, degree of hydrolysis 32% (WPC DH 32, 78% (w/w protein) Carbery Ingredients, Ballineen, Ireland), whey protein isolate hydrolysate, degree of hydrolysis 45% (WPI DH 45, 75% (w/w protein) Glanbia Nutritionals). The total protein content was 72.7g/100g powder. The protein matrix was supplemented with 2187mg/100g powder of milk-based calcium (Trucal™, Glanbia) and 57.3mg/100g powder vitamin D3 (cholecalciferol), flavoured and instantised to be dissolved in water.
  Other Names: MILK PROTEIN MATRIX (MPM)
  Arms: PROTEIN; PROTEIN+PHYSICAL ACTIVITY
Behavioral: PHYSICAL ACTIVITY — A structured, progressive programme of exercises using resistance exercise bands supervised by clinical therapists undertaken three times per week for 24 weeks of the intervention.
  Other Names: PA
  Arms: PROTEIN+PHYSICAL ACTIVITY

SUMMARY:
The focus is healthy ageing, i.e. delaying the deterioration in health status in older adults. Loss of lean tissue (skeletal muscle) mass, a process termed sarcopenia, or bone tissue mass, a process called osteopenia, is a consequence of aging per se, modified by nutrition and lifestyle behaviour.

The aim is to conduct a study of body composition, physical activity, muscle function and ability to undertake activities of daily living in older Irish men and women and to investigate the effect of a six month period of nutrient support, or nutrient plus physical activity on lean tissue mass and function and bone mass in men and women aged 50 to 70 years.

DETAILED DESCRIPTION:
Study Design: The study is a convenience population study and 6-month randomised control trial (RCT) of men and women age 55 to 70 years.

The study groups (n=60 per group) for the RCT are:

1. CON - a control group receiving a placebo nutrient support (per kg of body mass: 0.25g maltodextrin; energy ~ 160 kcal per day)
2. PRO - a nutrient group receiving a nutrient support (per kg of body mass: 0.33g milk protein + 0.25ug vitamin D + 10mg calcium; energy ~ 160 kcal per day)
3. PRO+PA - a nutrient group receiving a nutrient support (per kg of body mass: 0.33g milk protein + 0.25ug vitamin D + 10mg calcium; energy ~ 160 kcal per day) and engaging in a prescribed physical activity (PA).

Subject recruitment: Men and women, age 50 to 70 years, will be recruited through the UL Body Composition Study, by email advertisement, GP-exercise referral scheme, feature article(s) in the local media and word of mouth.

Requirement of the participants.

On entry each subject will undertake a preliminary assessment as follows:

i. medical history and examination by a qualified medical doctor ; ii. provide a blood and urine sample to be evaluated by a qualified medical doctor; iii. food intake evaluated by a qualified dietician; iv. whole body and segmental body composition analysis (DXA); v. habitual physical activity level (PAL) vi. measurement of muscle function and performance in simulated activities of daily living.

One month following the preliminary assessment subjects will be invited to participate in a 6 month intervention programme of nutrient or nutrient plus physical activity. Consenting subjects will be randomly assigned to one of the three study groups stated above.

Upon completion (6 months), subjects will be re-assessed as follows; i. provide a blood and urine sample; ii. whole body and segmental body composition analysis (DXA); iii. measurement of muscle function and performance in simulated activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Conducted by a medical doctor and based on Grieg et al. Age and Aging 1994:23:185-189 being defined as 'healthy' (i.e. 'disease-free') free-living and fully mobile older subjects capable of completing the 6-month intervention

Exclusion Criteria:

* Contraindication identified by medical doctor based on Grieg et al. Age and Aging 1994:23:185-189 definition of 'healthy' (i.e. 'disease-free') free-living and fully mobile older subjects capable of completing the 6-month intervention

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Body Lean Tissue Mass (LTM) | Change from baseline in Lean Tissue Mass at 6 months
  Body lean tissue mass measured by dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Bone Mineral Density | Change from baseline in Bone Mineral Density at 6 months
  Site specific (Lumbar Spine and Femoral Neck) bone mineral density measured by dual energy x-ray absorptiometry

OTHER OUTCOMES:
Maximal voluntary contraction (MVC) and rate of force development (RFD) of the knee extensors [Muscle Function] | Change from baseline in Muscle Function at 6 months
  Maximal voluntary contraction (MVC) in Nm (force in Newtons, distance in metres) torque of the knee extensors measured by ergometry will be used to assess Muscle Function.
Rate of force development (RFD) of the knee extensors [Muscle Function] | Change from baseline in Muscle Function at 6 months
  Rate of force development (RFD) in Nm/s (force in Newtons, distance in metres, time in seconds) torque of the knee extensors measured by ergometry will be used to assess Muscle Function.
Chair Rise Test [Activities of Daily Living] | Change from baseline in Activities of Daily Living at 6 months
  The number of completed Chair Rise (i.e. rise from a seated to a standing position) in 30 seconds will be used to assess Activities of Daily Living
Timed 1000m walk [Activities of Daily Living] | Change from baseline in Activities of Daily Living at 6 months
  The time (time in seconds) to complete 1000 metres (distance in metres) performed in a indoor track will be used to assess Activities of Daily Living

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jakeman, BSc MSc PhD, Principal Investigator — University of Limerick

REFERENCES:
- [Derived] Francis P, Mc Cormack W, Toomey C, Norton C, Saunders J, Kerin E, Lyons M, Jakeman P. Twelve weeks' progressive resistance training combined with protein supplementation beyond habitual intakes increases upper leg lean tissue mass, muscle strength and extended gait speed in healthy older women. Biogerontology. 2017 Dec;18(6):881-891. doi: 10.1007/s10522-016-9671-7. Epub 2016 Dec 8. PMID 27933408
- [Derived] Norton C, Toomey C, McCormack WG, Francis P, Saunders J, Kerin E, Jakeman P. Protein Supplementation at Breakfast and Lunch for 24 Weeks beyond Habitual Intakes Increases Whole-Body Lean Tissue Mass in Healthy Older Adults. J Nutr. 2016 Jan;146(1):65-9. doi: 10.3945/jn.115.219022. Epub 2015 Nov 18. PMID 26581685